CLINICAL TRIAL: NCT03269747
Title: Short Term Effect of Glucocorticoids on Brown Adipose Tissue Thermogenesis in Humans
Acronym: GlucoBAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EKNZ 2016-01859
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Brown Adipose Tissue
Keywords: glucocorticoids; brown adipose tissue; cold induced thermogenesis
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisone (Active Comparator): Prednisone 40 mg daily for 7 days
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator): Placebo daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — 2 tablets of Prednisone 20 Mg in the morning
  Arms: Prednisone
Drug: Placebo — 2 Placebo tablets in the morning
  Arms: Placebo

SUMMARY:
Interventional, Placebo controlled cross-over study to investigate the short-term effects of glucocorticoids (prednisone) on human brown adipose tissue.

DETAILED DESCRIPTION:
Active brown adipose tissue (BAT) has recently been unambiguously discovered in human adults. Active BAT increases energy expenditure and improves glucose tolerance. Pharmacological use of glucocorticoids (GCs) is widespread in clinical practice due to their high anti-inflammatory efficacy. While short-term administration even of high doses usually is well tolerated, long-term use of medium to high amounts of GCs leads to unfavorable metabolic changes, characterized by an increase in intra-abdominal fat mass, a decrease in muscle mass and insulin resistance.

In line with these well-known side-effects of GCs, several in vitro studies and animal models demonstrate an inhibiting effect of GCs on BAT thermogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* BMI between 19-27 kg/m2

Exclusion Criteria:

* Cold induced thermogenesis of less than 5% basal metabolic rate (determined during screening visit)
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* History of depressive disorder, anxiety disorder
* History of tuberculosis or latent infection
* Increased intraocular pressure
* History of peptic / gastrointestinal ulcer disease
* Concomitant medication: Non-steroidal anti-inflammatory drugs (NSAID), other glucocorticoids, diuretics, antihypertensives, fibrates or statins, metformin
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, diabetes mellitus),
* Hypersensitivity to cold (e.g. Raynaud Syndrome)
* Allergy to local anesthetic
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* Hypothyroidism without sufficient substitution
* Claustrophobia
* MRI incompatible implants
* Enrolment into another study using ionizing radiation within the previous 12 months.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Cold induced thermogenesis | at the end of each treatment period (day 7). Prednisone vs. Placebo
  : Increase in energy expenditure above resting metabolic rate in response to a mild cold stimulus determined by indirect calorimetry

SECONDARY OUTCOMES:
fat fraction of supraclavicular BAT | at the end of each treatment period (day 7). Prednisone vs. Placebo
  determined by MRI
volume of supraclavicular BAT | at the end of each treatment period (day 7). Prednisone vs. Placebo
  determined by MRI
cold stimulated FGD uptake in brown adipose tissue | at the end of each treatment period (day 7). Prednisone vs. Placebo
  determined as SUVmean by FDG-PET/CT
SUVmax in the supraclavicular adipose tissue depot | at the end of each treatment period (day 7). Prednisone vs. Placebo
  determined by FDG-PET/CT

OTHER OUTCOMES:
Glucose level before and after mild cold stimulus | at the end of each treatment period (day 7). Prednisone vs. Placebo
FGF21 level before and after mild cold stimulus | at the end of each treatment period (day 7). Prednisone vs. Placebo
Expression levels of genes involved in thermogenesis and white to brown adipose tissue transdifferentiation in supraclavicular adipose tissue. | at the end of each treatment period (day 7). Prednisone vs. Placebo

CONTACTS AND LOCATIONS:
Overall Officials: Matthias J Betz, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Department of Endocrinology, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Maushart CI, Sun W, Othman A, Ghosh A, Senn JR, Fischer JGW, Madoerin P, Loeliger RC, Benz RM, Takes M, Zech CJ, Chirindel A, Beuschlein F, Reincke M, Wild D, Bieri O, Zamboni N, Wolfrum C, Betz MJ. Effect of high-dose glucocorticoid treatment on human brown adipose tissue activity: a randomised, double-blinded, placebo-controlled cross-over trial in healthy men. EBioMedicine. 2023 Oct;96:104771. doi: 10.1016/j.ebiom.2023.104771. Epub 2023 Sep 4. PMID 37659283
- [Derived] Fischer JGW, Maushart CI, Becker AS, Muller J, Madoerin P, Chirindel A, Wild D, Ter Voert EEGW, Bieri O, Burger I, Betz MJ. Comparison of [18F]FDG PET/CT with magnetic resonance imaging for the assessment of human brown adipose tissue activity. EJNMMI Res. 2020 Jul 22;10(1):85. doi: 10.1186/s13550-020-00665-7. PMID 32699996